CLINICAL TRIAL: NCT00580593
Title: Pilot Placebo-Controlled Trial of Early Noninvasive Ventilation for ALS
Brief Title: Trial of Early Noninvasive Ventilation for Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Kirsten Gruis, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01NS55200
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; ALS; nocturnal noninvasive positive pressure ventilation; NIPPV; forced vital capacity; FVC
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: BiPAP® S/T System
- 2 (Sham Comparator)
  Interventions: Other: sham-NIPPV

INTERVENTIONS:
Device: BiPAP® S/T System — The BiPAP® S/T System is a NIPPV device that provides intermittent ventilatory assistance to people with difficulty breathing secondary to respiratory muscle weakness.
  Other Names: Noninvasive Positive Pressure Ventilation (NIPPV)
  Arms: 1
Other: sham-NIPPV — a sham-device
  Other Names: placebo
  Arms: 2

SUMMARY:
The goal of this trial is to determine the feasibility of conducting a randomized, double-blind, placebo-controlled trial of nocturnal noninvasive positive pressure ventilation in persons with amyotrophic lateral sclerosis with an forced vital capacity greater than or equal to 50 percent.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is an untreatable neurodegenerative disorder characterized by the progressive loss of motor neuron function. Respiratory failure is the most common cause of death in persons with ALS. Treatment of respiratory muscle weakness with nocturnal noninvasive positive pressure ventilation (NIPPV) when forced vital capacity (FVC) is less than 50 percent-but prior to the development of respiratory failure-has prolonged survival in observational studies. Despite the association of NIPPV use and survival, it is unknown whether earlier NIPPV treatment will benefit people with ALS. Also, no placebo-controlled studies of NIPPV treatment and people with ALS have been conducted.

The goals of the this trial are to assess the feasibility of conducting a prospective, randomized, double-blind, clinical trial of NIPPV versus control (sham) NIPPV in people with ALS who have a FVC greater than 50 percent, and to gain preliminary data on outcome effects.

In the trial, the investigators will test the following hypotheses: (1) People with ALS who have a FVC greater than 50 percent can tolerate active NIPPV and control NIPPV, and will find control NIPPV to be a believable treatment; (2) Initiation of active NIPPV in people with ALS who have a FVC greater than 50 percent will have better clinical outcomes with respect to measures of quality of life, rate of pulmonary function decline, and functional outcome; and (3) People with ALS who start active NIPPV early will have improved tolerance later when respiratory weakness has progressed. These aims will enable planning of a subsequent, large-scale and definitive clinical trial of early NIPPV (FVC greater than 50 percent) in people with ALS.

If the benefits of early NIPPV can be confirmed, then a new treatment may be established for this progressive, fatal disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Probable or possible ALS by El Escorial criteria
* If of child-bearing potential, has a negative urine or serum pregnancy test

Exclusion Criteria:

* FVC < 50% predicted for age
* Previous pneumothorax
* Bullous emphysema
* Requirement for oxygen
* Previous use of any positive pressure ventilation equipment (continuous positive airway pressure, or bilevel positive airway pressure)
* Current involvement in a clinical treatment trial
* Any unstable medical condition thought likely to interfere with participation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
NIPPV adherence, as summarized by weekly means and standard deviations of hours of use for the two groups (active-NIPPV and sham-NIPPV). Additionally the patients' belief as to which treatment they believed they had tried will be assessed. | every three months, for the duration of the disease or as long as the person with ALS is able to participate in the study.

SECONDARY OUTCOMES:
The SF-36 will be measured as a measure of quality of life. | at baseline and every three months
Pulmonary function tests including FVC will be measured. | at baseline and every three months
The ALS FRS will be used as a measure of functional outcome. | at baseline and every three months
The BDI/TDI (baseline and transition dyspnea indexes). | at baseline and every three months
Tolerance to standard NIPPV treatment during the observational phase of the study (after FVC has fallen below 50%) will also be summarized by weekly means and standard deviations of hours of use. | at baseline and every three months

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Gruis, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Jacobs TL, Brown DL, Baek J, Migda EM, Funckes T, Gruis KL. Trial of early noninvasive ventilation for ALS: A pilot placebo-controlled study. Neurology. 2016 Nov 1;87(18):1878-1883. doi: 10.1212/WNL.0000000000003158. Epub 2016 Aug 31. PMID 27581221